CLINICAL TRIAL: NCT00996073
Title: A Prospective, Multicenter, Randomized, Open-Label, Controlled Study Evaluating Safety and Preliminary Efficacy of NeoFuse When Combined With MasterGraft Matrix in Subjects Undergoing Lumbar Interbody Fusion With Instrumentation
Brief Title: Safety and Preliminary Efficacy Study of NeoFuse in Subjects Requiring Lumbar Interbody Fusion
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mesoblast, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MSB-SF003
Record Dates: First submitted 2009-10-09; First posted 2009-10-16 (Estimated); Last update posted 2020-06-29 (Actual); Status verified 2020-06

CONDITIONS: Degenerative Disc Disease; Degenerative Spondylolisthesis; Spinal Stenosis
Keywords: Degenerative disc disease; Spondylolisthesis; Spinal stenosis; Stem cells; Adult Stem Cells; Spinal Fusion; Lumbar Spinal Fusion; TLIF; PLIF; Mesoblast
MeSH Terms: conditions — Intervertebral Disc Degeneration; Spinal Stenosis; Spondylolisthesis | interventions — Transplantation, Autologous; Spinal Fusion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Autograft (Active Comparator): Lumbar Interbody Fusion with Autograft
  Interventions: Biological: Lumbar Interbody Fusion with Autograft
- Low Dose (Experimental): Lumbar Interbody Fusion with NeoFuse-Low Dose
  Interventions: Biological: Lumbar Interbody Fusion with NeoFuse
- High Dose (Experimental): Lumbar Interbody Fusion with NeoFuse-High Dose
  Interventions: Biological: Lumbar Interbody Fusion with NeoFuse

INTERVENTIONS:
Biological: Lumbar Interbody Fusion with Autograft — Single Dose Autograft Surgical Implantation
  Other Names: Spinal Fusion; Control
  Arms: Autograft
Biological: Lumbar Interbody Fusion with NeoFuse — Single Dose NeoFuse Surgical Implantation
  Other Names: Spinal Fusion; Stem Cells
  Arms: Low Dose
Biological: Lumbar Interbody Fusion with NeoFuse — Single Dose NeoFuse Surgical Implantation
  Other Names: Spinal Fusion; Stem Cells
  Arms: High Dose

SUMMARY:
The purpose of this study is to evaluate the safety and preliminary efficacy of NeoFuse in subjects with a diagnosis of degenerative disc disease (DDD) in 1 or 2 adjacent vertebral levels between L1 and S1. All subjects in this study will undergo interbody fusion via Transforaminal Lumbar Interbody Fusion (TLIF) or Posterior Lumbar Interbody Fusion (PLIF) procedures with Food and Drug Administration (FDA) approved/cleared supplemental posterior instrumentation.

DETAILED DESCRIPTION:
This is a prospective, multicenter, randomized, open-label controlled Phase 2 study designed to evaluate the safety and preliminary efficacy of adult, allogeneic mesenchymal precursor cells (MPCs) combined with MasterGraft Matrix when compared to use of autologous iliac crest bone graft in the lumbar interbody fusion site in subjects requiring 1 or 2 level interbody fusion procedure with instrumentation. All subjects in this study will undergo a 1 or 2-level (2 or 3 vertebrae) interbody fusion with supplemental posterior instrumentation.

After the screening and surgical visits, each subject will be evaluated clinically and radiographically within 3 days and 30 days after surgery, and at 3, 6, 9, 12, 24, and 36 months after surgery.

Subjects will be evaluated at the same time points for safety.

ELIGIBILITY:
Inclusion Criteria:

1. Male or females at least 18 years of age, but not older than 70.
2. Have the ability to understand the requirements of the study, to provide written informed consent, and to comply with the study protocol.
3. Have the ability to understand and provide written authorization for the use and disclosure of personal health information (PHI) [per Health Insurance Portability and Accountability Act (HIPAA) privacy ruling in the US].
4. Have a documented symptomatic diagnosis of DDD at L1-S1 with or without stenosis and with or without up to and including Grade II degenerative spondylolisthesis.
5. Have clinical symptoms of neurogenic claudication.
6. Have failed 6 months of non-operative low back pain management.
7. Are candidates for posterior lumbar interbody fusion in combination with posterior pedicle screw stabilization and require surgery at a 1 or 2 adjacent vertebral levels between L1 and S1.
8. Have a stable screening electrocardiogram (ECG), as determined by the investigator that would not preclude surgery.

Exclusion Criteria:

1. Female subjects who are pregnant or nursing, or women planning to become pregnant during the first year (12 months) following surgery.

   * Male subjects with partners of childbearing potential must agree to use adequate contraception (barrier method or abstinence) from the time of surgery and for a period of at least 1 year after surgery.
2. Have a current or prior history within the last 3 years of neoplasm (excluding basal cell carcinoma) and/or any active neoplasm within the last 24 months, prior to screening.
3. Have osteoporosis as defined by a DEXA T score of ≤ -3.0 or a history of fragility fractures or other significant bone disease contraindicating the use of spinal instrumentation.
4. Have a documented medical history or radiographic evidence of a metabolic bone disease or other condition which would negatively impact the bone healing process.
5. Have a positive screen for human immunodeficiency virus (HIV) antibodies.
6. Have had treatment with any investigational therapy or device within 6 months of study surgery and/or plans to participate in any other allogeneic stem cell/progenitor cell therapy trial during the 3-year follow-up period.
7. Have been a recipient of prior stem cell/progenitor cell therapy for spinal fusion surgery.
8. Have a body mass index (BMI) > 35.
9. Have 20% or greater anti-human leukocyte antigen (HLA) antibody titer and/or has antibody specificities to donor HLA antigens.
10. Are transient or has been treated in the last 6 months before enrollment for alcohol and/or drug abuse in an inpatient substance abuse program.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-09; Primary Completion 2012-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
To determine the overall safety of NeoFuse plus carrier using physical examinations, vital signs, treatment emergent adverse events (TEAEs), and the results of clinical lab tests (hematology, serum chemistry, inflammation, and immunology). | 3 years

SECONDARY OUTCOMES:
To evaluate the overall fusion success with NeoFuse plus carrier compared to autograft using CT scans and x-ray of the involved lumbar spine levels and assess the change in outcomes (ODI, SF-36, and WPAI) and pain (VAS)at the 12-month follow-up visit. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Roger Brown, Study Director — Senior Vice President of Musculoskeletal Repair
Locations (5):
- United States (5):
  - The Spine Institute, Santa Monica, California
  - Denver Spine, Greenwood Village, Colorado
  - Rocky Mountain Associates in Orthopedic Medicine, P.C., Loveland, Colorado
  - Fort Wayne Orthopaedics, Fort Wayne, Indiana
  - Central Texas Spine Institute, Austin, Texas

REFERENCES:
- See also: The Sponsor's web site — http://www.mesoblast.com